CLINICAL TRIAL: NCT06484764
Title: Validate the Feasibility and Safety of the Robot System by Comparing the CT-fluoroscopy Guidance Versus CT-guided Freehand Needle Biopsy in Participants With Suspected Thoracic or Abdominal Lesions in a Randomized Controlled Trial
Brief Title: Validate the Safety and Feasibility of the CT-guided Interventional Robot in Percutaneous Biopsy Procedure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Tongji Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Wuhan United Imaging Healthcare-Surgical Technology Co., Ltd. Wuhan, China (Unknown)
Responsible Party: Principal Investigator, Haipeng Yu, Professor, Chief Physician, Tianjin Medical University Cancer Institute and Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: ZRIR-003-22-01
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Abdominal Cancer; Thoracic Cancer
Keywords: Image guided biopsy; Robot-assisted method

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-fluoroscopy guided robot-assisted percutaneous needle biopsy group (Experimental): Remote controlled, CT-fluoroscopy guided, robot-assisted biopsy procedure of thoracic and abdominal lesions
  Interventions: Procedure: CT-fluoroscopy guided robot-assisted biopsy of thoracic and abdominal lesions
- Freehand needle biopsy group under the CT guidance (Active Comparator): Freehand CT-guided percutaneous needle biopsy of thoracic and abdominal lesions
  Interventions: Procedure: Freehand CT-guided percutaneous needle biopsy of thoracic and abdominal lesions

INTERVENTIONS:
Procedure: CT-fluoroscopy guided robot-assisted biopsy of thoracic and abdominal lesions — During the procedure, the participant first undergoes a CT scan the radiologist plans the needle trajectory based on the registered preoperative CECT (contrast-enhanced computed tomography
  ) and intraoperative CT. After the participant is manually sterilised and given local anaesthesia, the radiologist will remotely control the robot to finish the needle insertion process under the CT-fluoroscopy guidance and simultaneously adjust the angular needle if necessary. The radiologist confirms whether the needle has reached the target area by CT-fluoroscopy image.
  Arms: CT-fluoroscopy guided robot-assisted percutaneous needle biopsy group
Procedure: Freehand CT-guided percutaneous needle biopsy of thoracic and abdominal lesions — Radiologists following the current clinical practice guidance to finish the freehand biopsy procedure under the CT guidance.
  Arms: Freehand needle biopsy group under the CT guidance

SUMMARY:
This multicenter, randomized controlled trial aims to investigate whether the interventional robot can be well and safely used for percutaneous needle biopsy compared with the freehand needle biopsy method under CT guidance in patients with suspected thoracic or abdominal lesions. The robot allows radiologists to remotely control the needle insertion process under the CT-fluoroscopy guidance. The main questions it aims to answer are:

1. Whether the robot-assisted needle biopsy method can decrease patient radiation exposure during the biopsy procedure.
2. Whether the robot-assisted needle biopsy method can improve the success rate for radiologists to insert the needle into the target lesions area without additional needle adjustment
3. Whether the robot-assisted needle biopsy method can decrease the patient's complication occurrence rate
4. Whether the robot-assisted needle biopsy method can decrease the time from the beginning to the end of needle insertion.

All the participants with suspected thoracic and abdominal lesions will be randomly assigned to the study group or control group.

Participants in the study group will receive a robot-assisted biopsy procedure under the CT-fluoroscopy guidance.

Participants in the control group will receive a freehand needle biopsy under the CT guidance.

DETAILED DESCRIPTION:
Cancer has become the second main death reason among Chinese residents. According to the latest global cancer burden data for 2020 released by the International Agency for Research on Cancer (IARC) of the World Health Organization, there were 4.57 million new cases of cancer and more than 3 million deaths in China in 2020, accounting for 23.7% and 30.2% respectively of the total number of global cancer incidence and deaths in 2020. Early detection and early treatment have become crucial to reducing cancer incidence and mortality. Image-guided percutaneous needle biopsy has been an important and established method for tumour treatment and diagnosis. More specifically, physicians under CT, MRI (magnetic resonance imaging) or ultrasound guidance manually insert a puncture needle into the target area of the soft tissue lesion for biopsy. However, the image-guidance freehand biopsy method still faces the following challenges:

1. Lack of real-time and accurate information during the needle insertion process, including puncture force, needle deformation, soft tissue deformation, and needle arrival position;
2. Multiple scans during the puncture are needed to determine whether the needle has successfully reached the target area, which leads to prolonged operation time, easily induces complications and increases the radiation dose to the physicians.
3. The accuracy of needle insertion is highly affected by the patient's respiration movement causing the multi-directional nonlinear displacement and deformation of tissues and organs (movement, rotation, etc.), resulting in the drift of the tumour position. Eventually, it is difficult for radiologists to insert the target position, resulting in false negative results of biopsy or procedure failure.
4. The physiological trembling of the radiologist's hand will reduce the accuracy of puncture, and even lead to complications such as bleeding and pneumothorax
5. Percutaneous puncture procedure is highly dependent on the ability and experience of radiologists.

Here, the investigators aim to evaluate whether the robot-assisted needle biopsy method can solve these challenges by comparing the safety and feasibility of robotic-assisted percutaneous needle biopsy with freehand needle biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Participants have suspected thoracic or abdomen lesions.
* Participants need to receive CT-guided non-vascular percutaneous biopsy procedure
* Lesion size ≥ 10 mm that confirmed by radiologists through the preoperative CT.

Exclusion Criteria:

* Participants with uncorrectable coagulopathy, infectious lesions in the planned needle trajectory path, pulmonary echinococcosis considered on CT imaging, patients who need mechanical ventilation, hepatic alveolar echinococcosis, coma or other diseases that the investigators think not suitable for joining the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
One-time puncture success rate | The same day of the procedure
  The criteria for successful one-time puncture were as follows: the operator judged that the needle had reached the target area without any needle withdrawal or needle direction change during the puncture time that from the needle tip penetrated the skin to the time that needle reached to the target area.
  The one-time puncture success rate = number of participants with one-time puncture success (study group or control group) / total number of subjects in the (study group or control group)*100%

SECONDARY OUTCOMES:
The number of needle adjustments | The same day of the procedure
  The number will be counted when the needle tip angle was altered or needle retreat during puncture procedure.
Procedure time | The same day of the procedure
  Time from the patient was positioned to the arrival at the target area that confirmed by CT imaging.
Puncture time | The same day of the procedure
  Time from the needle tip at the skin entry point to the puncture was completed.
Radiation exposure dose to the patient | The same day of the procedure
  Total radiation dose received by patient during the procedure
Complication rate | Three days after the procedure
  The proportion of patients with complications in the two groups. Complications including pneumothorax, pneumothorax, hemoptysis, bleeding and other adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Haipeng, PhD,MD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital; Nan Wang, PhD,MD, Principal Investigator — Tongji Hospital; Bin Xiong, MD, PhD, Principal Investigator — First Clinical Affiliation of Guangzhou Medical University
Locations (3):
- China (3):
  - First Clinical Affiliation of Guangzhou Medical University, Guangzhou
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Tongji Hospital of Huazhong University of Science and Technology, Wuhan